CLINICAL TRIAL: NCT00124332
Title: Randomized, Multicenter, Double-Blind, Placebo-Controlled, Two-Arm Parallel Group Trial of Rimonabant 20-mg od, for Inhibition of Atherosclerosis Progression Assessed by IVUS (IntraVascular UltraSounds), in Overweight Patients With Clustering Risk Factors
Brief Title: STRADIVARIUS (Strategy To Reduce Atherosclerosis Development InVolving Administration of Rimonabant - the Intravascular Ultrasound Study)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC5827
Record Dates: First submitted 2005-07-26; First posted 2005-07-27 (Estimated); Last update posted 2009-04-20 (Estimated); Status verified 2009-04

CONDITIONS: Coronary Atherosclerosis
MeSH Terms: conditions — Coronary Artery Disease | interventions — Rimonabant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: Rimonabant (SR141716)
Drug: Placebo

SUMMARY:
The purpose of this study is to determine if rimonabant 20 mg once daily (od) administered during 18-20 months will reduce progression of coronary atherosclerosis as assessed by intravascular ultrasound (IVUS) when administered on top of standard behavioral and pharmacological therapy given as needed, in patients with abdominal obesity associated with current smoking and/or metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Written and signed informed consent
* Indication for coronary angiography
* Abdominal obesity defined by waist circumference > 88 cm in women or > 102 cm in men
* At least one of the two following conditions: *a) Metabolic syndrome as defined by the presence of at least two of the following additional risk factors: 1. Triglyceride level >= 150 mg/dL (1.69 mmol/L); 2. HDL cholesterol < 40 mg/dL (1.03 mmol/L) [men] or 50 mg/dL (1.28 mmol/L) [women]; 3. Fasting glucose >= 110 mg/dL (6.1 mmol/L); 4. High blood pressure (>= 140 mmHg systolic and/or >= 90 mmHg diastolic) at Screening visit, or current treatment by anti-hypertensive medication; *b) Currently smoking (> 10 cigarettes /day) and willing to stop
* Angiographic evidence of coronary heart disease as defined by at least 1 lesion in a native coronary artery that has >= 20% reduction in lumen diameter by angiographic visual estimation
* Presence of at least one coronary artery complying with the definition of "target vessel" for IVUS assessment
* Acceptation of the Baseline IVUS tape by the IVUS Core Laboratory

Exclusion Criteria:

* Age < 18 years
* Pregnant or breast-feeding women
* History of very low-calorie diet or surgical procedures for weight loss (eg, stomach stapling, bypass) within 6 months prior to screening visit
* Obesity of known endocrine origin
* Uncontrolled diabetes with HBA1c >10%
* Presence of any severe medical or psychological condition, that in the opinion of the Investigator would compromise the subject's safety or successful participation in the study
* Severe congestive heart failure (New York Heart Association [NYHA] Class III or IV)
* Clinically significant heart disease which in the opinion of the Investigator is likely to require coronary artery bypass graft (CABG), percutaneous coronary intervention (PCI), cardiac transplantation, surgical repair and/or replacement during the course of the study
* Angioplasty of a non-qualifying artery which is considered at high risk of acute complication or restenosis, during baseline catheterization
* >50% reduction in lumen diameter of the left main coronary artery by visual angiographic estimation
* Recent ST-elevation myocardial infarction (MI) <= 72 hours prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 839 (Actual)
Dates: Start 2005-01; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
change from baseline in percent atheroma volume (PAV) | Month 18 visit

SECONDARY OUTCOMES:
change from baseline in normalized total atheroma volume (TAV) | Month 18 visit

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (9):
- The Cleveland Clinic Foundation, Cleveland, Ohio, United States
- sanofi-aventis, Australia, Macquarie Park, Australia
- sanofi-aventis, Belgium, Diegem, Belgium
- Sanofi-Aventis Administrative Office, Laval, Canada
- sanofi-aventis, France, Paris, France
- sanofi-aventis Italy, Milan, Italy
- sanofi-aventis, Netherlands, Gouda, Netherlands
- sanofi-aventis Poland, Warsaw, Poland
- sanofi-aventis Spain, Barcelona, Spain

REFERENCES:
- [Result] Nissen SE, Nicholls SJ, Wolski K, Rodes-Cabau J, Cannon CP, Deanfield JE, Despres JP, Kastelein JJ, Steinhubl SR, Kapadia S, Yasin M, Ruzyllo W, Gaudin C, Job B, Hu B, Bhatt DL, Lincoff AM, Tuzcu EM; STRADIVARIUS Investigators. Effect of rimonabant on progression of atherosclerosis in patients with abdominal obesity and coronary artery disease: the STRADIVARIUS randomized controlled trial. JAMA. 2008 Apr 2;299(13):1547-60. doi: 10.1001/jama.299.13.1547. Epub 2008 Apr 1. PMID 18387931